CLINICAL TRIAL: NCT02829320
Title: A 24-week, Phase III, Open-label, Non-comparative, Multi-center Study to Evaluate Efficacy and Safety of GSK1278863 in Japanese Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease Who Are Not Taking Erythropoiesis Stimulating Agents
Brief Title: Efficacy and Safety Study of GSK1278863 in Japanese Hemodialysis Subjects With Anemia Associated With Chronic Kidney Disease Who Are Not Taking Erythropoiesis Stimulating Agents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204716
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Anaemia
Keywords: efficacy; hemodialysis (HD); hemoglobin (Hgb); erythropoiesis-stimulating agents (ESAs); GSK1278863
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1278863 (Experimental): Subjects will receive GSK1278863 once daily orally at a starting dose of 4 milligrams (mg) on Day 1, and continued until the day of Week 4. From Weeks 4 to 24, interruption of treatment or dose adjustments will be made within the maintenance dose range of 1 mg to 24 mg according to the dose adjustment algorithm to achieve and/or maintain Hgb within the target range (10.0 to 12.0 g/dL) based on the Hgb value measured every 4 weeks. Dose changes will be made every 4 weeks. Iron replacement therapy will be given according to the standard starting criteria.
  Interventions: Drug: GSK1278863; Drug: Iron

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863 will be provided as round, standard biconvex, white film coated tablets containing 1 mg, 2 mg, 4 mg or 6 mg of GSK1278863 as active ingredient.
Drug: Iron — Subjects will receive supplemental iron therapy if ferritin is <=100 ng/mL and TSAT is <=20%. The investigator (or subinvestigator) will choose the route of administration and dose of prescription iron.

SUMMARY:
This 24-week, Phase 3, open-label, non-comparative, multicentre study aims to evaluate the efficacy and safety of GSK1278863 in Japanese hemodialysis (HD) patients with renal anemia not using erythropoiesis-stimulating agents (ESAs). The primary objective is to evaluate the initial response to GSK1278863 measured by hemoglobin (Hgb) levels in HD patients not using ESAs enrolled in this study. The study is designed to evaluate the appropriateness of the starting dose of GSK1278863 and of the GSK1278863 dose adjustment regimen to achieve or maintain the target Hgb levels. This study will consist of a 4-week screening period, a 24-week treatment period (4-week fixed-dose period and a 20-week dose adjustment period), and a 2- to 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age (at the time of informed consent): >=20 years
* Dialysis: Patients on hemodialysis (HD) or hemodiafiltration (HDF)
* Use of any erythropoiesis stimulating agent (ESA): Newly started dialysis (Dialysis newly started <12 weeks before screening): Patients not using ESAs after the start of dialysis; Maintenance dialysis (Dialysis started >=12 weeks before screening): Patients not using ESAs within 8 weeks before screening (including interruption of ESA therapy)
* Hemoglobin (Hgb): >=8.0 to <10.0 g/dL (measured using a point-of-care Hgb measurement device at the study site on Day 1)
* Iron parameter: Ferritin >100 nanograms (ng)/milliliter (mL) or transferrin saturation (TSAT) >20% (at screening only)
* Gender (at screening only): Female or male.

A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test for females of reproductive potential [FRP] only), not breastfeeding, and at least one of the following conditions applies:

* Females of non-reproductive potential defined as: Pre-menopausal with one of the following and no plans to utilise assisted reproductive techniques (example [e.g.], in vitro fertilisation or donor embryo transfer): documented bilateral tubal ligation or salpingectomy; documented hysteroscopic tube occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; documented bilateral oophorectomy
* Post-menopausal defined as females 60 years of age or older or In females <60 years of age, 12 months of spontaneous amenorrhea (In questionable cases, a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause is confirmatory [the reference values are provided separately]). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

Females of reproductive potential who agree to follow one of the options listed in the "GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential" from 28 days before the first dose of study treatment until completion of the follow-up visit.

* Informed consent: Subjects who can provide written informed consent to the study, involving compliance with the requirements and patient responsibilities stated in the consent form and the protocol.

Exclusion Criteria:

CKD related criteria

* Kidney transplant: Planned living kidney transplant during the study period Anemia-related criteria
* Aplasia: History of bone marrow aplasia or pure red cell aplasia
* Other causes of anemia: Pernicious anemia, thalassaemia, sickle cell disease, or myelodysplastic syndrome
* Gastrointestinal bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant gastrointestinal bleeding within 8 weeks before screening or during a period from screening to Day 1.

Cardiovascular disease-related criteria

* History of myocardial infarction, acute coronary syndrome, stroke or transient ischemic attack: Diagnosed within 8 weeks before screening or during a period from screening to Day 1.
* Heart failure: Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system
* Corrected QT interval (QTc) (at screening only): QTc >500 milliseconds (msec), or QTc >530 msec in subject with bundle branch block. Note: Corrected QT interval using Bazett's formula (QTcB) (machine-read or manually) will be used.

Other disease-related criteria

* Liver disease (if any of the following occurs):

  * Alanine transaminase (ALT) >2x upper limit of normal (ULN)
  * Bilirubin >1.5xULN (If bilirubin fractions are measured and direct bilirubin is <35%, isolated bilirubin >1.5xULN will be acceptable.)
  * Current unstable active liver or biliary disease (generally defined by the onset of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, persistent jaundice, or cirrhosis). Note: The only exception is squamous cell or basal cell carcinoma of the skin that has been definitively treated >=8 weeks before screening.
* Malignancy: History of malignancy within the two years prior to screening, known complex kidney cyst >3 centimeters (cm) (II F, III or IV based on the Bosniak classification) or currently receiving treatment for cancer. Note: The only exception is squamous cell or basal cell carcinoma of the skin that has been definitively treated >=8 weeks before screening.

Concomitant medications and other study treatment-related criteria

* Iron medication: Planned use of any intravenous iron during the screening period or from Day 1 to Week 4.

Note:

* Patients on oral iron may be enrolled if the iron dose regimen is unchanged during the screening period and from Day 1 to Week 4.
* Patients on anti-hyperphosphatemia medication containing iron (e.g., ferric citrate hydrate) for at least 12 weeks before screening may be enrolled if the medication is continued during the screening and from Day 1 to Week 4.

  * Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to any excipients in the investigational product
  * Drugs and dietary supplements: Current use of prohibited prescription drugs, non-prescription drugs, or dietary supplements or planned use of any of these drugs during the study period (prohibited drugs: strong cytochrome P450 (CYP)2C8 inducers and inhibitors)
  * Exposure to any other investigational product: Use of an investigational product within the past 30 days or five half lives of that investigational product (whichever is longer).
  * Prior treatment with GSK1278863: Prior treatment with GSK1278863 for >30 days General health-related criteria
  * Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Japan (13):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20062

REFERENCES:
- [Background] Tsubakihara Y, Akizawa T, Nangaku M, Onoue T, Yonekawa T, Matsushita H, Endo Y, Cobitz A. A 24-Week Anemia Correction Study of Daprodustat in Japanese Dialysis Patients. Ther Apher Dial. 2020 Apr;24(2):108-114. doi: 10.1111/1744-9987.12962. Epub 2019 Aug 13. PMID 31306555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 24-week, Phase 3, open-label, non-comparative, multicenter study to evaluate the efficacy and safety of GSK1278863 in Japanese hemodialysis participants with renal anemia not using Erythropoiesis Stimulating Agents. The study was conducted at 18 centers in Japan from 08-Aug-2016 to 17-Oct-2017.
Pre-assignment Details: A total of 36 participants were screened and 8 failed screening because of not meeting eligibility criteria (7) and withdrawal by participants (1). The remaining 28 participants were enrolled in this study. This study consisted of a 4-week screening period, a 24-week treatment period and a 2 to 4-week follow-up period.
Groups:
- All Participants: Participants with newly started dialysis (dialysis newly started <12 weeks before screening) or with maintenance dialysis (dialysis started >=12 weeks before screening) received GSK1278863 orally once daily initially at 4 milligram (mg) for 4 weeks from Day 1. Subsequently, participants received GSK1278863 orally once a day according to a pre-defined study treatment dose adjustment algorithm to achieve or maintain hemoglobin (Hgb) within the target range (10.0-12.0 grams per deciliter [g/dL]). In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 nanogram per milliliter (ng/mL) and transferrin saturation (TSAT) is <=20%.
Period: Overall Study
Arm/Group | All Participants
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All Treated Subjects
Groups:
- All Participants: Participants with newly started dialysis (dialysis newly started <12 weeks before screening) or with maintenance dialysis (dialysis started >=12 weeks before screening) received GSK1278863 orally once daily initially at 4 mg for 4 weeks from Day 1. Subsequently, participants received GSK1278863 orally once a day according to a pre-defined study treatment dose adjustment algorithm to achieve or maintain Hgb within the target range (10.0-12.0 g/dL). In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Treated Subjects
  Years | 62.5 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Treated Subjects
  Participants
    Female | 3
    Male | 25
Race/Ethnicity, Customized [Number; unit: Count of Participants] — Population: All Treated Subjects
  Count of Participants
    Asian - Japanese Heritage | 28
Dialysis Status [Count of Participants; unit: Participants] — Dialysis newly started < 12 weeks before screening was considered as Newly started dialysis. Dialysis started >= 12 weeks before screening was considered as Maintenance dialysis.
  Participants
    Newly started dialysis | 11
    Maintenance dialysis | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hgb at Week 4
Description: Blood samples were collected from participants for measurement of Hgb values. The Baseline value was the latest pre-dose assessment. Change from Baseline at Week 4 was calculated by subtracting Baseline value from the post-dose visit value. The analysis was performed on All Treated Subjects Population which comprised of all participants who received at least one dose of GSK1278863.
Time Frame: Baseline and Week 4
Population: All Treated Subjects Population
Measure: Mean (95% Confidence Interval); unit: G/dL
Arm/Group | All Participants
Number analyzed (Participants) | 28
G/dL | 0.79 [0.53 to 1.05]

2. Primary Outcome: Number of Participants by Hgb Change From Baseline Category at Week 4
Description: Blood samples were collected from participants for measurement of Hgb values. The Baseline value was the latest pre-dose assessment. Change from Baseline at Week 4 was calculated by subtracting Baseline value from the post-dose visit value. The change in Hgb at Week 4 was classified into different categories (i.e., <=-2.0, >-2.0 to -1.0, >-1.0 to 0, >0 to 1.0, >1.0 to 2.0, and >2 g/dL), and the number of participants in each category were summarized.
Time Frame: Baseline and Week 4
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants
  <= -2.0 | 0
  > -2.0 to -1.0 | 0
  > -1.0 to 0 | 4
  > 0 to 1.0 | 13
  > 1.0 to 2.0 | 11
  > 2.0 | 0

3. Secondary Outcome: Hgb Values at the Indicated Time Points
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: G/dL
Arm/Group | All Participants
Number analyzed (Participants) | 28
G/dL
  Day 1 | 9.10 (0.696)
  Week 4 | 9.90 (0.907)
  Week 8 | 10.76 (0.957)
  Week 12 | 11.09 (1.117)
  Week 16 | 11.38 (1.286)
  Week 20 | 11.34 (1.169)
  Week 24 | 11.12 (1.210)

4. Secondary Outcome: Change From Baseline in Hgb at the Indicated Time Points
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The Baseline value was the latest pre-dose assessment. Change from Baseline at indicated time-points was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: G/dL
Arm/Group | All Participants
Number analyzed (Participants) | 28
G/dL
  Week 4 | 0.79 (0.673)
  Week 8 | 1.66 (0.773)
  Week 12 | 1.98 (0.984)
  Week 16 | 2.28 (1.248)
  Week 20 | 2.24 (1.174)
  Week 24 | 2.01 (1.121)

5. Secondary Outcome: Number of Participants Who Had Hgb Level Within the Target Range (10.0-12.0 g/dL)
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The number of participants with Hgb withinthe target range (10.0 to 12.0 g/dL) at each assessment visit was summarized.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants
  Day 1, within range | 3
  Week 4, within range | 13
  Week 8, within range | 20
  Week 12, within range | 18
  Week 16, within range | 17
  Week 20, within range | 20
  Week 24, within range | 23

6. Secondary Outcome: Time to Reach the Lower Target Hgb Level (10.0 g/dL)
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. Participants who could not reach lower target were regarded as censored. The time (in days) to reach the lower target Hgb level (10.0 g/dL) was summarized using 25th percentile (P25), median, and 75th percentile (P75) by Kaplan-Meier method.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 28
Days | 57.0 [29.0 to 57.0]

7. Secondary Outcome: Number of Participants Who Had Hgb Level of Less Than 7.5 g/dL
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The number of participants who had Hgb level of less than 7.5 g/dL were summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits were included.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants | 0

8. Secondary Outcome: Number of Participants Who Had Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The number of participants who had Hgb increase of more than 2.0 g/dL over any 4 weeks were summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits were included.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants | 1

9. Secondary Outcome: Number of Participants Who Had Hgb Level of More Than 13.0 g/dL
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The number of participants who had Hgb level of more than 13.0 g/dL were summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits were included.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants | 3

10. Secondary Outcome: Number of Episodes of Achieving Hgb Level of More Than 13.0 g/dL
Description: Blood samples were collected from participants for measurement of Hgb values at indicated time points. Hgb was evaluated using Hgb analyzer. The number of episodes in participants who had Hgb level of more than 13.0 g/dL were summarized. On-therapy Hgb values observed in both scheduled and unscheduled visits were included.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Number; unit: Episodes
Arm/Group | All Participants
Number analyzed (Participants) | 28
Episodes | 7

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to 4 Hours (AUC [0-4]) of GSK1278863
Description: Blood samples were collected to evaluate AUC (0-4) at 1, 2, 3 and 4 hours post dose at Weeks 12 and 24. Pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis. PK Population consisted of all participants who received GSK1278863 with the PK samples collected and analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indiates data was not available. Geometric coefficient of variation could not be calculated when number of participant was equal to 1.
Time Frame: 1, 2, 3 and 4 hours post dose at Weeks 12 and 24
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Groups:
- GSK1278863 1 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 1 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 2 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 2 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 4 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 4 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 6 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 6 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 8 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 8 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 12 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 12 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
- GSK1278863 18 mg: Participants received GSK1278863 orally once daily initially at 4 mg from Day 1 in 4-week fixed-dose period. Participants received GSK1278863 18 mg orally at specified visits just before collecting the PK samples. As PK samples were collected more than once, participants might be included in more than one arm. In participants taking oral iron before the study, their iron dose was not changed during the fixed-dose period. Supplemental iron therapy was administered if ferritin is <=100 ng/mL and TSAT is <=20%.
Arm/Group | GSK1278863 1 mg | GSK1278863 2 mg | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 12 mg | GSK1278863 18 mg
Number analyzed (Participants) | 1 | 12 | 22 | 13 | 3 | 1 | 1
Hour*nanogram per milliliter (h*ng/mL)
  AUC (0-4), Week 12, n=0,4,14,8,1,0,0: number analyzed (Participants) | 0 | 4 | 14 | 8 | 1 | 0 | 0
  AUC (0-4), Week 12, n=0,4,14,8,1,0,0 |  | 25.7228 (289.9) | 95.1319 (111.9) | 200.6036 (62.9) | 233.3933 (NA) — The dispersion was not calculated because of n=1 |  |
  AUC (0-4), Week 24, n=1,8,8,5,2,1,1: number analyzed (Participants) | 1 | 8 | 8 | 5 | 2 | 1 | 1
  AUC (0-4), Week 24, n=1,8,8,5,2,1,1 | 43.3100 (NA) — The dispersion was not calculated because of n=1 | 33.8941 (230.9) | 86.3702 (58.9) | 133.3020 (50.9) | 437.0983 (18.7) | 749.4583 (NA) — The dispersion was not calculated because of n=1 | 126.2883 (NA) — The dispersion was not calculated because of n=1
  AUC (0-4), All, n=1,12,22,13,3,1,1 | 43.3100 (NA) — The dispersion was not calculated because of n=1 | 30.9164 (225.3) | 91.8474 (91.1) | 171.4229 (60.8) | 354.6083 (40.0) | 749.4583 (NA) — The dispersion was not calculated because of n=1 | 126.2883 (NA) — The dispersion was not calculated because of n=1

12. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK1278863
Description: Blood samples were collected to evaluate Cmax at 1, 2, 3 and 4 hours post dose at Weeks 12 and 24. PK parameters were calculated by standard non-compartmental analysis. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indiates data was not available. Geometric coefficient of variation could not be calculated when number of participant was equal to 1.
Time Frame: 1, 2, 3 and 4 hours post dose at Weeks 12 and 24
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK1278863 1 mg | GSK1278863 2 mg | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 12 mg | GSK1278863 18 mg
Number analyzed (Participants) | 1 | 12 | 22 | 13 | 3 | 1 | 1
ng/mL
  Cmax, Week 12, n=0,4,14,8,1,0,0: number analyzed (Participants) | 0 | 4 | 14 | 8 | 1 | 0 | 0
  Cmax, Week 12, n=0,4,14,8,1,0,0 |  | 13.9578 (340.6) | 57.6572 (81.2) | 122.9883 (56.9) | 179.0000 (NA) — The dispersion was not calculated because of n=1 |  |
  Cmax, Week 24, n=1,8,8,5,2,1,1: number analyzed (Participants) | 1 | 8 | 8 | 5 | 2 | 1 | 1
  Cmax, Week 24, n=1,8,8,5,2,1,1 | 27.5000 (NA) — The dispersion was not calculated because of n=1 | 18.3448 (202.3) | 44.8853 (49.8) | 100.2261 (41.3) | 202.9384 (3.5) | 311.0000 (NA) — The dispersion was not calculated because of n=1 | 93.4000 (NA) — The dispersion was not calculated because of n=1
  Cmax, All, n=1,12,22,13,3,1,1 | 27.5000 (NA) — The dispersion was not calculated because of n=1 | 16.7474 (217.4) | 52.6391 (70.4) | 113.6784 (50.4) | 194.6229 (7.7) | 311.0000 (NA) — The dispersion was not calculated because of n=1 | 93.4000 (NA) — The dispersion was not calculated because of n=1

13. Secondary Outcome: Monthly Average Dose of Intravenous (IV) Iron During the Treatment Period
Description: Records of on-therapy iron medication were used to calculate average quarterly IV iron dose. Quarter 1 = (Randomization Date - Treatment Start Date at Week 12 - 1 [day]). Quarter 2 = (Treatment Start Date at Week 12 - Study Treatment Stop Date). Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: Mg
Arm/Group | All Participants
Number analyzed (Participants) | 28
Mg
  Quarter 1; n= 3: number analyzed (Participants) | 3
  Quarter 1; n= 3 | 231.61 (99.916)
  Quarter 2; n= 4: number analyzed (Participants) | 4
  Quarter 2; n= 4 | 217.19 (86.529)

14. Secondary Outcome: Number of Participants Who Used Iron During the Treatment Period
Description: The number of participants who used iron (both IV and oral iron) during the treatment period were summarized.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants
  Oral iron | 9
  Intravenous iron | 4
  Any iron medication | 12

15. Secondary Outcome: Change From Baseline in Ferritin
Description: Blood samples were collected from participants for measurement of serum ferritin at indicated time points. The Baseline value was the latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: Microgram per liter (µg/L)
Arm/Group | All Participants
Number analyzed (Participants) | 28
Microgram per liter (µg/L)
  Week 4 | -80.11 (51.826)
  Week 12 | -126.29 (120.382)
  Week 24 | -107.03 (143.048)

16. Secondary Outcome: Percent Change From Baseline in TSAT
Description: Blood samples were collected from participants for measurement of TSAT at indicated time points. The Baseline value was the latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1).
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of transferrin
Arm/Group | All Participants
Number analyzed (Participants) | 28
Percentage of transferrin
  Week 4 | -23.06 [-32.43 to -12.38]
  Week 12 | -15.31 [-33.79 to 8.32]
  Week 24 | -10.07 [-25.49 to 8.55]

17. Secondary Outcome: Percent Change From Baseline in Hepcidin
Description: Blood samples were collected from participants for measurement of hepcidin at indicated time points. The Baseline value was the latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1). If a laboratory value had a non-detectable level reported in the database, where the numeric value was missing, the value was not included in a summary. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of hepcidin
Arm/Group | All Participants
Number analyzed (Participants) | 28
Percentage of hepcidin
  Week 4, n=26: number analyzed (Participants) | 26
  Week 4, n=26 | -64.78 [-71.34 to -56.71]
  Week 12, n=22: number analyzed (Participants) | 22
  Week 12, n=22 | -61.74 [-74.51 to -42.57]
  Week 24, n=21: number analyzed (Participants) | 21
  Week 24, n=21 | -55.67 [-72.52 to -28.47]

18. Secondary Outcome: Change From Baseline in Serum Iron
Description: Blood samples were collected from participants for measurement of serum iron at indicated time points. The Baseline value was the latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | All Participants
Number analyzed (Participants) | 28
Micromoles per liter (µmol/L)
  Week 4 | -0.8123 (4.92624)
  Week 12 | 2.0916 (10.74722)
  Week 24 | 1.4584 (7.72121)

19. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity (TIBC)
Description: Blood samples were collected from participants for measurement of TIBC at indicated time points. The Baseline value was the latest pre-dose assessment. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Week 24
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | All Participants
Number analyzed (Participants) | 28
umol/L
  Week 4 | 8.5904 (4.93732)
  Week 12 | 10.8611 (6.32355)
  Week 24 | 9.3388 (9.92131)

20. Secondary Outcome: Dose Level of GSK1278863 at Indicated Time Points
Description: Dose adjustment algorithm was used which was based on Hgb values at scheduled visits. Hgb values measured at unscheduled visits were not included. Mean dose during Week 12 to 24 is the average of dose at Weeks 12, 16, and 20.
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Median (Full Range); unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 28
mg
  Day 1 | 4.0 [4 to 4]
  Week 4 | 4.0 [2 to 6]
  Week 8 | 4.0 [2 to 8]
  Week 12 | 4.0 [0 to 8]
  Week 16 | 4.0 [0 to 12]
  Week 20 | 4.0 [0 to 18]
  Week 12 to 24 | 4.00 [0.0 to 12.7]

21. Secondary Outcome: Number of Participants With Frequency of Dose Adjustments
Description: Dose adjustment algorithm was used which was based on Hgb values at scheduled visits. Hgb values measured at unscheduled visits were not included. For dose adjustments frequency, the number of participants were provided by the number of dose adjustments (i.e. zero, one, two, three, four, and five or more).
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 28
Participants
  Any dose adjustments | 21
  Number of dose adjustments=0 | 7
  Number of dose adjustments=1 | 9
  Number of dose adjustments=2 | 7
  Number of dose adjustments=3 | 4
  Number of dose adjustments=4 | 1
  Number of dose adjustments=5 or more | 0

22. Secondary Outcome: Duration of Treatment Interruption Due to Hgb >13 g/dL
Description: Hgb values were used for making decision of treatment interruption. On-therapy Hgb values observed in both scheduled and unscheduled visits were counted. Participants who have no treatment interruption due to Hgb >13.0 g/dL are not included
Time Frame: Up to Week 24
Population: All Treated Subjects Population
Measure: Median (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 3
Days | 84 [28 to 84]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study treatment (Day 1) until Week 24.
Description: On-treatment SAEs and non-serious AEs are reported for All Treated Subjects Population.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 3/28
Other Adverse Events (participants affected / at risk) | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=28)
Shunt occlusion (Injury, poisoning and procedural complications) | 2 (3)
Device dislocation (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=28)
Nasopharyngitis (Infections and infestations) | 9 (10)
Infected dermal cyst (Infections and infestations) | 2 (3)
Shunt stenosis (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02829320/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02829320/SAP_001.pdf